CLINICAL TRIAL: NCT04426266
Title: Psychological Effects of the COVID-19 Pandemic on the Hungarian Adult Population
Status: Completed | Type: Observational
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: PSZ-002
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-06

CONDITIONS: Questionnaire Designs; COVID-19 Pandemic; Psychological Stress; Coping Skills; Two-Item Generalised Anxiety Disorder Scale; Patient Health Questionnaire Anxiety and Depression Scale; Health Status Index; Subjective Health Complaint; Mood
MeSH Terms: conditions — COVID-19; Stress, Psychological; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to explore the psychological effects of the COVID-19 pandemic among Hungarian adults with the use of an anonymous online questionnaire that consists of 65 items. With these results it will possible to identify coping strategies that can help Hungarian adults to deal with the difficulties arising from the pandemic.

DETAILED DESCRIPTION:
Planned course of the project:

1. We make the questionnaire using Google Forms.
2. The link of the online questionnaire is sent to three public groups via the social media website Facebook.
3. By clicking on the sent link, all participants are able to read information about the project and about the consent to participate in it. Then the participant will be able to give consent to participate in the project. After giving consent, the participant will be able to start filling out the questionnaire. If the participant indicates that he/she does not want to give consent to the study, the website will indicate that the participation of him/her has ended in the project.
4. Anonymous answers will be automatically saved.
5. The participants will be given code numbers based on the order in which they filled out the questionnaire.
6. The data will be analysed by the researchers. For a participant, completing the online questionnaire takes approximately 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

The participant must have access to the internet and to the social media website Facebook.

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult Hungarian
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
sociodemopraphic factors | 5 months
  6 items - age, sex, city of residence, marital status, level of education, employment status
perceived stress | 5 months
  Perceived Stress Scale (PSS), 10 items about thoughts and feelings that characterize a person's perception of stress
level of anxiety | 5 months
  The General Anxiety Disorder Assessment GAD-2, 2 items to examine the level of anxiety
self-reported health state | 5 months
  EQ5D-VAS, 1 item to examine health status
number of complaints | 5 months
  Self-administered inventory of complaints (Hungarian questionnaire), 20 items to measure number of complaints.
strategies in coping with stressful situations | 5 months
  Shortened (Hungarian) version of the Ways of Coping Questionnaire (WOC), 22 items to measure cognitive or behavioral strategies in coping with stressful situations
psychological effects of the coronavirus pandemic on the participants' mood and ways of coping with difficulties arising from the pandemic | 5 months
  psychological effects of the coronavirus pandemic on the participants' mood and ways of coping with difficulties arising from the pandemic, 2 open-ended questions (not obligatory to answer) in connection with psychological effects of the coronavirus pandemic (its effects on the participants' mood and ways of coping with difficulties arising from the pandemic).
level of depression | 5 months
  The Patient Health Questionnaire PHQ-2, 2 items to examine the level of depression

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Kemény, Prof. Dr., Principal Investigator — University of Szeged, Department of Dermatology and Allergology
Locations (1):
- University of Szeged Department of Dermatology and Allergology, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xiao C. A Novel Approach of Consultation on 2019 Novel Coronavirus (COVID-19)-Related Psychological and Mental Problems: Structured Letter Therapy. Psychiatry Investig. 2020 Feb;17(2):175-176. doi: 10.30773/pi.2020.0047. Epub 2020 Feb 25. No abstract available. PMID 32093461
- [Background] Ho CS, Chee CY, Ho RC. Mental Health Strategies to Combat the Psychological Impact of Coronavirus Disease 2019 (COVID-19) Beyond Paranoia and Panic. Ann Acad Med Singap. 2020 Mar 16;49(3):155-160. No abstract available. PMID 32200399
- [Background] Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, Ho RC. Immediate Psychological Responses and Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19) Epidemic among the General Population in China. Int J Environ Res Public Health. 2020 Mar 6;17(5):1729. doi: 10.3390/ijerph17051729. PMID 32155789